CLINICAL TRIAL: NCT04449666
Title: Investigation of the Relationship Between Hippocampal Volume and Memory Functions in in Patients With Aneurysmal Subarachnoid Hemorrhage (aSAH)
Brief Title: Hippocampal Volume and Memory Functions in Aneurysmal Subarachnoid Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: SAB-VOL
Record Dates: First submitted 2020-06-18; First posted 2020-06-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neurologic Disorder; Subarachnoid Hemorrhage, Aneurysmal
Keywords: Neurological rehabilitation; Hippocampal volume; Memory deficits
MeSH Terms: conditions — Nervous System Diseases; Subarachnoid Hemorrhage; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: Patients undergoing neurological rehabilitation after aneurysmal subarachnoid hemorrhage
  Interventions: Diagnostic Test: Neuropsychological assessment and structural MRI
- Control group: Healthy adults controlled for age, gender and educational status
  Interventions: Diagnostic Test: Neuropsychological assessment and structural MRI

INTERVENTIONS:
Diagnostic Test: Neuropsychological assessment and structural MRI — Complex neuropsychological assessment testing attentional and memory functions. Additionally, a structural MRI is measured.

SUMMARY:
Neuropsychological and functional long-term consequences of subarachnoid hemorrhages (SAH) represent a great challenge, since sometimes considerable cognitive deficits occur without evidence of substantial brain damage. In this study, we want to examine if the frequently observed memory deficits are associated with hippocampal atrophy.

DETAILED DESCRIPTION:
Long-term or even permanent neuropsychological impairments are frequently observed after aneurysmal subarachnoid hemorrhages (aSAH). Among the most common impairments after aSAH are memory deficits. Volumetric MRI studies suggest an association of memory dysfunctions with temporal atrophy, especially of the hippocampus. In a previous study, 77 patients with good or moderate clinical outcome after aSAH were examined one year after discharge (Bendel et al., 2006). Temporomesial atrophy was detected without direct brain damage, e.g. by secondary ischemia. Due to the effects of complex cognitive impairments on the quality of life and participation in social and professional life, this relationship will be examined in more detail in the planned study. Specifically, we will investigate to what extent the frequently observed discrepancy between severe memory impairment and normal structural imaging results (no focal lesions in temporomesial areas) is due to hippocampal atrophy. In contrast to Bender and colleagues, this question will be investigated in the acute phase of the disease, immediately after admission to inpatient neurological rehabilitation.

Over a period of 24 months, 29 neurological rehabilitation patients with aSAH (Hunt & Hess grade I and II) are going to be included. Within the first week (day 1 to 7) after study enrollment, a native MRI examination (without contrast agent) is performed, in which a high-resolution 3D-MPRAGE sequence (T1 weighting) is measured in the sagittal plane. After checking the data quality of the 3D-MPRAGE sequence, especially with regard to its suitability for hippocampal volume determination, a comprehensive neuropsychological examination is performed, in which specific memory and attentional functions are tested.

ELIGIBILITY:
Inclusion Criteria:

* neurological rehabilitation patients in phase B - D
* at minimum eight weeks after disease onset
* aneurysmal subarachnoid hemorrhage (Hunt & Hess grade I or II)
* written consent from the patient's legal representative
* exclusion of pregnancy

Exclusion Criteria:

* insufficient cardiorespiratory stability
* previous brain damage
* mental disorders (dementia, depression)
* colonization with multi-resistant pathogens
* MRI contraindications
* claustrophobia
* weight > 120 kg

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: neurological rehabilitation patients with aneurysmal subarachnoid hemorrhage (Hunt & Hess grade I or II)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Changed hippocampal volume in aSAB | 2 weeks
  Hypothesis: patients have smaller hippocampal volume than healthy control subjects. For the hippocampal volume a structural MRI scan (3D-MPRAGE) is obtained

SECONDARY OUTCOMES:
Changed memory function in aSAB | 2 weeks
  Hypothesis: patients have lower scores in the Visual and Verbal memory test (VVM) than healthy control subjects.
Influence of the type of therapy on the hippocampal volume | 2 weeks
  Hypothesis: hippocampal volumes differ between aSAH patients with surgical or endovascular treatment.
Influence of the lesion site on the hippocampal volume | 2 weeks
  Hypothesis: there are no differences between ispi- and contralateral hippocampal volumes
Interrater reliability | 2 weeks
  Hypothesis: It is expected that there will be no difference in the ratings of hippocampal volume between two independent raters.
Changed intracranial volume in aSAB | 2 weeks
  Hypothesis: patients have smaller intracranial volume than healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Rollnik, MD, Study Director — BDH-Clinic Hessisch Oldendorf; Melanie Boltzmann, PhD, Principal Investigator — BDH-Clinic Hessisch Oldendorf
Locations (1):
- BDH-Clinic Hessisch Oldendorf, Hessisch Oldendorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Period of availability begins when results are published, at the earliest in Dec 2022
Access Criteria: IPD can be obtained from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Bendel P, Koivisto T, Hanninen T, Kolehmainen A, Kononen M, Hurskainen H, Pennanen C, Vanninen R. Subarachnoid hemorrhage is followed by temporomesial volume loss: MRI volumetric study. Neurology. 2006 Aug 22;67(4):575-82. doi: 10.1212/01.wnl.0000230221.95670.bf. PMID 16924007